CLINICAL TRIAL: NCT04713202
Title: Prospective Assessment of Patients With Neuroendocrine Tumors and Current or Prior History of Carcinoid Syndrome or Diarrhea Undergoing Peptide Receptor Radionuclide Therapy With or Without Telotristat Ethyl (NET-PACS Trial) Big Ten Cancer Research Consortium BTCRC-GI19-400
Brief Title: Prospective Assessment of Patients With Neuroendocrine Tumors and Current or Prior History of Carcinoid Syndrome or Diarrhea Undergoing Peptide Receptor Radionuclide Therapy With or Without Telotristat Ethyl
Acronym: NET-PACS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funder decision
Sponsor: Chandrikha Chandrasekhara (Other)
Responsible Party: Sponsor-Investigator, Chandrikha Chandrasekhara, Clinical Assistant Professor of Internal Medicine - Hematology, Oncology and Blood and Marrow Transplantation, Big Ten Cancer Research Consortium
Organization: Big Ten Cancer Research Consortium (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: BTCRC-GI19-400
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Neuroendocrine Tumors; Carcinoid Syndrome; Diarrhea
MeSH Terms: conditions — Neuroendocrine Tumors; Serotonin Syndrome; Diarrhea | interventions — telotristat ethyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Telotristat Ethyl + PRRT (Experimental): Telotristat ethyl, 250 mg, PO, three times daily, continuous.
  + Peptide Receptor Radionuclide Therapy(PRRT) every 8 weeks
  Interventions: Drug: Telotristat ethyl; Drug: Peptide Receptor Radionuclide Therapy
- Placebo + PRRT (Placebo Comparator): Placebo, PO, three times daily, continuous.
  + Peptide Receptor Radionuclide Therapy(PRRT) every 8 weeks
  Interventions: Drug: Peptide Receptor Radionuclide Therapy; Other: Placebo

INTERVENTIONS:
Drug: Telotristat ethyl — Telotristat Ethyl, 250mg
  Arms: Telotristat Ethyl + PRRT
Drug: Peptide Receptor Radionuclide Therapy — Peptide Receptor Radionuclide Therapy
  Other Names: PRRT
Other: Placebo — Placebo
  Arms: Placebo + PRRT

SUMMARY:
The NET-PACS trial is a Prospective Assessment of patients with neuroendocrine tumors and current or prior history of Carcinoid Syndrome or diarrhea undergoing peptide receptor radionuclide therapy with or without telotristat ethyl. The main goal of the study is to demonstrate the feasibility of serial in-depth assessment of patients with neuroendocrine tumors and current or prior history of carcinoid syndrome or diarrhea undergoing treatment with PRRT using telotristat ethyl compared to placebo. We aim to report and describe from a patient's perspective the multi-faceted impact of carcinoid syndrome in patients with NETs and the changes on treatment while getting PRRT using telotristat ethyl compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Males and females, aged 18 and older
* Histologically-confirmed neuroendocrine tumor (GI or other primary)
* Presence of somatostatin receptors as by either Ga-68 dotatate imaging or Octreoscan or comparable method, which is a requirement for PRRT (Lutathera ®). Disease does not need to be measurable per RECIST since it is not uncommon to have non-target lesions but not meet criteria for RECIST as long as presence of somatostatin receptors can be demonstrated. NOTE: Patients undergoing other types of PRRT would not be eligible for this clinical trial.
* Eligible for treatment with PRRT (Lutathera®) according to institutional practice and product label.
* Patient with current or prior history of symptomatic carcinoid syndrome or carcinoid diarrhea as per investigator assessment. Note: prior history and current controlled carcinoid patients are eligible.
* Demonstrate adequate organ function as defined in the protocol; all screening labs to be obtained within 28 days prior to registration.
* Life expectancy greater than 12 weeks as per investigator opinion
* ECOG performance status 0-2
* Women of childbearing potential (WOCBP) must have a negative pregnancy test (urine or serum βhCG) within 7 days prior to study registration. If a urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. See the protocol for WOCBP definition.

Exclusion Criteria:

* Surgery, radiotherapy, within 4 weeks; chemotherapy, or other investigational therapy within 2 weeks prior to study registration, or 5 half-lives of a drug, whichever is shorter.
* Uncontrolled congestive heart failure prior to study registration. Patients can be considered eligible if the disease is controlled at the date of randomization.
* Subject with another significant medical, psychiatric, or surgical conditions, currently uncontrolled by treatment, which may interfere with completion of the study as per investigator opinion.
* Women of childbearing potential (WOCBP), must agree to use appropriate method(s) of contraception. Women are considered to be of childbearing potential unless are surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause).
* WOCBP must agree to use appropriate method(s) of contraception from the time of informed consent until 7 months post-treatment completion. Complete abstinence is also an acceptable form of contraception.
* Men who are sexually active with WOCBP must agree to use appropriate method(s) of contraception from the first dose of study drug until 4 months post-treatment completion. Complete abstinence is also an acceptable form of contraception.
* Telotristat ethyl tablets contain lactose as an excipient. Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency, or glucose-galactose malabsorption should not take telotristat ethyl.
* Concomitant medications: Any other herbal or alternative medicines being used as an anti-cancer treatment are not allowed. NOTE: if patient is receiving a drug that is a CYP3A4 substrate, strongly consider switching to an alternate drug if possible. The latter is more of a recommendation, not an exclusion criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
FACT-QS global QoL Score | From enrollment until completion of study therapy or subject withdrawal, up to six months
  Feasibility of in-depth assessment of changes and improvement on treatment in patients undergoing treatment as determined by FACT-CS global QoL with PRRT using telotristat ethyl compared to placebo. The FACT-CS global QoL is the primary endpoint. Scores will be derived using FACIT guidelines and will range from 0 to 12 with higher scores denoting a better level of functioning.
  A repeated measures ANOVA will be applied and statistical significance of fixed effects of treatment arm, time and treatment arm by time interaction will be assessed using a Wilks' Lambda Approximate F test.

SECONDARY OUTCOMES:
To describe and report from a patient's perspective the multi-faceted impact of carcinoid syndrome in patients with NETs and the changes on treatment while getting PRRT using telotristat ethyl compared to placebo. | From enrollment until completion of study therapy or subject withdrawal, up to six months
  Linear mixed effects regression model will be utilized to describe longitudinal changes in QoL as measured by the identified FACT-CS scales. Fixed effects for treatment arm, time and treatment arm by time interaction along with a random effect to account for the longitudinally correlated nature of repeated questionnaire measurements will be included. Graphical plots of the estimated mean and associated 95% confidence intervals by time point in the study will be produced.
ATo report changes in patient reported outcomes (PRO) in the diarrhea domain in patients undergoing PRRT receiving telotristat ethyl versus placebo. | From enrollment until completion of study therapy or subject withdrawal, up to six months
  Linear mixed effects regression model will be utilized to describe longitudinal changes in QoL Diarrhea domain as measured by the identified FACT-CS scales. Fixed effects for treatment arm, time and treatment arm by time interaction along with a random effect to account for the longitudinally correlated nature of repeated questionnaire measurements will be included. Graphical plots of the estimated mean and associated 95% confidence intervals by time point in the study will be produced.
To report changes in patient reported outcomes (PRO) in the flushing domain in patients undergoing PRRT receiving telotristat ethyl versus placebo. | From enrollment until completion of study therapy or subject withdrawal, up to six months
  Linear mixed effects regression model will be utilized to describe longitudinal changes in QoL as measured by the identified FACT-CS scales in the flushing domain. Fixed effects for treatment arm, time and treatment arm by time interaction along with a random effect to account for the longitudinally correlated nature of repeated questionnaire measurements will be included. Graphical plots of the estimated mean and associated 95% confidence intervals by time point in the study will be produced.
To estimate the need of rescue short-acting somatostatin receptor antagonist in patients undergoing PRRT receiving telotristat ethyl versus placebo. | From enrollment until completion of study therapy or subject withdrawal, up to six months
  Linear mixed effects regression model will be utilized to describe longitudinal changes in frequency of rescue short acting somatostatin receptor antagonist use. Fixed effects for treatment arm, time and treatment arm by time interaction along with a random effect to account for the longitudinally correlated nature of repeated questionnaire measurements will be included. Graphical plots of the estimated mean and associated 95% confidence intervals by time point in the study will be produced.
To estimate the weight-gain in patients undergoing PRRT receiving telotristat ethyl versus placebo. | From enrollment until completion of study therapy or subject withdrawal, up to six months
  Linear mixed effects regression model will be utilized to describe longitudinal changes in weight. Fixed effects for treatment arm, time and treatment arm by time interaction along with a random effect to account for the longitudinally correlated nature of repeated questionnaire measurements will be included. Graphical plots of the estimated mean and associated 95% confidence intervals by time point in the study will be produced.
To estimate the changes in bowel movement frequency and/or consistency in patients undergoing PRRT receiving telotristat ethyl versus placebo. | From enrollment until completion of study therapy or subject withdrawal, up to six months
  Linear mixed effects regression model will be utilized to describe longitudinal changes in frequency and/or changes in consistency of bowel movements. Fixed effects for treatment arm, time and treatment arm by time interaction along with a random effect to account for the longitudinally correlated nature of repeated questionnaire measurements will be included. Graphical plots of the estimated mean and associated 95% confidence intervals by time point in the study will be produced.

CONTACTS AND LOCATIONS:
Overall Officials: Chandrikha Chandrasekharan, MD, Principal Investigator — University of Iowa; Al B Benson, MD, Study Chair — Northwestern University
Locations (1):
- University of Iowa Hospital and Clinics, Iowa City, Iowa, United States